CLINICAL TRIAL: NCT05922618
Title: PEMFS in Patients With CRPS-I of the Foot and Ankle: a Randomized Controlled Trial
Brief Title: Pulsed Electromagnetic Fields (PEMFS) in Complex Regional Pain Syndrome Type i (CRPS-I) of the Foot (PeCFoA)
Acronym: (PeCFoA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PeCFoA
Record Dates: First submitted 2023-06-08; First posted 2023-06-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Pain, Joint; Complex Regional Pain Syndromes; Ankle Disease; Foot Diseases
Keywords: Complex Regional Pain Syndromes; foot; ankle
MeSH Terms: conditions — Arthralgia; Complex Regional Pain Syndromes; Foot Diseases

STUDY DESIGN:
Intervention Model Description: Spontaneous, prospective, randomized study with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-ONE group (Experimental): The group will undergo home biophysical treatment with I-ONE® therapy (experimental group) for 4 hours/day for 60 days. Patients will follow standard rehabilitation treatment: patients will perform active and active-assisted range of motion (ROM) recovery exercises and stretching exercises for 30 minutes per day, for 6 weeks.
  Interventions: Device: I-One
- Exercise group (No Intervention): The group, not subjected to biophysical therapy, will be controls. Patients will follow standard rehabilitation treatment: patients will perform active and active-assisted ROM recovery exercises and stretching exercises for 30 minutes per day, for 6 weeks.

INTERVENTIONS:
Device: I-One — I-ONE® is a medical device certified by the Ministry of Health as a Medical Device (risk class II A) for the treatment of inflammatory and degenerative tissue pathologies. The device consists of a signal generator and an applicator, called a solenoid. The solenoid will be placed on the joint, not necessarily in direct contact with the skin. The device works with a rechargeable battery and is equipped with an hour counter to assess patient compliance.
  Treatment with I-ONE® therapy will start within 3-7 days of recruitment, will last 6 hours a day and will be maintained for 60 days. The treatment will be carried out at home and the device will be delivered directly to the patient's home by courier.
  Other Names: I-One, IGEA, Italy
  Arms: I-ONE group

SUMMARY:
The investigators hypothesize that the association of I-ONE® therapy with standard rehabilitation treatment can optimize the clinical and functional recovery of patients with pulsed electromagnetic fields (PEMFs) (I-ONE® therapy) of the foot or ankle.

DETAILED DESCRIPTION:
Study design; spontaneous, prospective, randomized study with control group.

Purpose of the study:

evaluate the functional clinical improvement of the foot/ankle joint with algodystrophic pathology following a standard rehabilitation treatment and home biophysical treatment and local biophysical stimulation with I-ONE® therapy (IGEA SpA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type I CRPS according to the Budapest criteria (table 1)
* Type I CRPS involving the ankle or foot
* Onset of CRPS type I up to a maximum of 3 years after the symptomatic event
* Pain on visual analog scale (VAS) scale quantified as intensity at least ≥ 5 at recruitment
* Pharmacological treatment with first infusion cycle of neridronate

Exclusion Criteria:

* Neurological pathologies (stroke, degenerative, traumatic pathologies)
* Local neurological impairment (type II CRPS), confirmed by a conduction test or similar
* Cardiac pacemaker, treatment site malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with allodynia | Change from baseline at 3 months
  • Clinical assessment of allodynia (tested as pain by lightly stroking with a small brush (end of a cotton swab: dichotomic present/absent response)
Number of participants with allodynia | Change from baseline at 6 months
  • Clinical assessment of allodynia (tested as pain by lightly stroking with a small brush (end of a cotton swab: dichotomic present/absent response)
Number of participants with allodynia | Change from baseline at 12 months
  • Clinical assessment of allodynia (tested as pain by lightly stroking with a small brush (end of a cotton swab: dichotomic present/absent response)
Number of participants with hyperalgesia | Change from baseline at 3 months
  Clinical evaluation of hyperalgesia (defined as a pin prick-evoked stimulus perceived as something more painful or longer than the duration of the stimulus in the affected limb compared to the contralateral limb: dichotomic present/absent response)
Number of participants with hyperalgesia | Change from baseline at 12 months
  Clinical evaluation of hyperalgesia (defined as a pin prick-evoked stimulus perceived as something more painful or longer than the duration of the stimulus in the affected limb compared to the contralateral limb: dichotomic present/absent response)
Rate of edema | Change from baseline at 3 months
  • Local edema (score 0=none, 1=mild, 2=moderate, 3=severe, at the level of the ankle and midfoot, by direct comparison with the healthy contralateral limb)
Rate of edema | Change from baseline at 6 months
  • Local edema (score 0=none, 1=mild, 2=moderate, 3=severe, at the level of the ankle and midfoot, by direct comparison with the healthy contralateral limb)
Rate of edema | Change from baseline at 12 months
  • Local edema (score 0=none, 1=mild, 2=moderate, 3=severe, at the level of the ankle and midfoot, by direct comparison with the healthy contralateral limb)
Pain at movement | Change from baseline at 3 months
  Pain evoked by passive movement (ankle and toe joints for foot involvement) was rated as 0=none, 1=mild, 2=moderate, 3=severe, by direct comparison with the healthy contralateral limb)
Pain at movement | Change from baseline at 6 months
  Pain evoked by passive movement (ankle and toe joints for foot involvement) was rated as 0=none, 1=mild, 2=moderate, 3=severe, by direct comparison with the healthy contralateral limb)
Pain at movement | Change from baseline at 12 months
  Pain evoked by passive movement (ankle and toe joints for foot involvement) was rated as 0=none, 1=mild, 2=moderate, 3=severe, by direct comparison with the healthy contralateral limb)
Pain intensity | Change from baseline at 3 months
  Visual Analogue Scale (VAS): the Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Pain intensity | Change from baseline at 6 months
  Visual Analogue Scale (VAS): the Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Pain intensity | Change from baseline at 12 months
  Visual Analogue Scale (VAS): the Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Pain intensity | at 12 months
  Visual Analogue Scale (VAS): the Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

SECONDARY OUTCOMES:
Evaluate a better recovery of joint functionality | Change from baseline at 3 months
  •• American Foot & Ankle Score (AOFAS): scores range from 0 to 100, with healthy ankles receiving 100 points.
Evaluate a better recovery of joint functionality | Change from baseline at 6 months
  •• American Foot & Ankle Score (AOFAS): scores range from 0 to 100, with healthy ankles receiving 100 points.
Evaluate a better recovery of joint functionality | Change from baseline at 12 months
  •• American Foot & Ankle Score (AOFAS): scores range from 0 to 100, with healthy ankles receiving 100 points.
Self-reporting measure of pain | Change from baseline at 3 months
  McGill Pain Questionnaire: scores range from 0 (no pain) to 78 (severe pain)
Self-reporting measure of pain | Change from baseline at 6 months
  McGill Pain Questionnaire: scores range from 0 (no pain) to 78 (severe pain)
Self-reporting measure of pain | Change from baseline at 12 months
  McGill Pain Questionnaire: scores range from 0 (no pain) to 78 (severe pain)
Number of participants taking medications | Change from baseline at 3 months
  • Assessment report for Non-Steroidal Anti-Inflammatory Drugs
Number of participants taking medications | Change from baseline at 6 months
  • Assessment report for Non-Steroidal Anti-Inflammatory Drugs
Number of participants taking medications | Change from baseline at 12 months
  • Assessment report for Non-Steroidal Anti-Inflammatory Drugs
patient assessment of pain and limitations of activity | Change from baseline at 3 months
  he Roles and Maudsley score is a subjective 4-point patient assessment of pain and limitations of activity (1 = excellent result with no symptoms following treatment; 2 = significant improvement from pre-treatment; 3 = patient somewhat improved; 4 = poor, symptoms identical or worse than pre- treatment)
patient assessment of pain and limitations of activity | Change from baseline at 6 months
  he Roles and Maudsley score is a subjective 4-point patient assessment of pain and limitations of activity (1 = excellent result with no symptoms following treatment; 2 = significant improvement from pre-treatment; 3 = patient somewhat improved; 4 = poor, symptoms identical or worse than pre- treatment)
patient assessment of pain and limitations of activity | Change from baseline at 12 months
  he Roles and Maudsley score is a subjective 4-point patient assessment of pain and limitations of activity (1 = excellent result with no symptoms following treatment; 2 = significant improvement from pre-treatment; 3 = patient somewhat improved; 4 = poor, symptoms identical or worse than pre- treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Angela Notarnicola, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adravanti P, Nicoletti S, Setti S, Ampollini A, de Girolamo L. Effect of pulsed electromagnetic field therapy in patients undergoing total knee arthroplasty: a randomised controlled trial. Int Orthop. 2014 Feb;38(2):397-403. doi: 10.1007/s00264-013-2216-7. Epub 2013 Dec 20. PMID 24352823
- [Background] Benazzo F, Cadossi M, Cavani F, Fini M, Giavaresi G, Setti S, Cadossi R, Giardino R. Cartilage repair with osteochondral autografts in sheep: effect of biophysical stimulation with pulsed electromagnetic fields. J Orthop Res. 2008 May;26(5):631-42. doi: 10.1002/jor.20530. PMID 18176941
- [Background] Benazzo F, Zanon G, Pederzini L, Modonesi F, Cardile C, Falez F, Ciolli L, La Cava F, Giannini S, Buda R, Setti S, Caruso G, Massari L. Effects of biophysical stimulation in patients undergoing arthroscopic reconstruction of anterior cruciate ligament: prospective, randomized and double blind study. Knee Surg Sports Traumatol Arthrosc. 2008 Jun;16(6):595-601. doi: 10.1007/s00167-008-0519-9. Epub 2008 Apr 2. PMID 18385980
- [Background] Bigoni M, Sacerdote P, Turati M, Franchi S, Gandolla M, Gaddi D, Moretti S, Munegato D, Augusti CA, Bresciani E, Omeljaniuk RJ, Locatelli V, Torsello A. Acute and late changes in intraarticular cytokine levels following anterior cruciate ligament injury. J Orthop Res. 2013 Feb;31(2):315-21. doi: 10.1002/jor.22208. Epub 2012 Aug 6. PMID 22886741
- [Background] de Girolamo L, Stanco D, Galliera E, Vigano M, Colombini A, Setti S, Vianello E, Corsi Romanelli MM, Sansone V. Low frequency pulsed electromagnetic field affects proliferation, tissue-specific gene expression, and cytokines release of human tendon cells. Cell Biochem Biophys. 2013 Jul;66(3):697-708. doi: 10.1007/s12013-013-9514-y. PMID 23345006
- [Background] de Girolamo L, Vigano M, Galliera E, Stanco D, Setti S, Marazzi MG, Thiebat G, Corsi Romanelli MM, Sansone V. In vitro functional response of human tendon cells to different dosages of low-frequency pulsed electromagnetic field. Knee Surg Sports Traumatol Arthrosc. 2015 Nov;23(11):3443-53. doi: 10.1007/s00167-014-3143-x. Epub 2014 Jun 24. PMID 24957914
- [Background] De Mattei M, Pasello M, Pellati A, Stabellini G, Massari L, Gemmati D, Caruso A. Effects of electromagnetic fields on proteoglycan metabolism of bovine articular cartilage explants. Connect Tissue Res. 2003;44(3-4):154-9. PMID 14504035
- [Background] De Mattei M, Pellati A, Pasello M, Ongaro A, Setti S, Massari L, Gemmati D, Caruso A. Effects of physical stimulation with electromagnetic field and insulin growth factor-I treatment on proteoglycan synthesis of bovine articular cartilage. Osteoarthritis Cartilage. 2004 Oct;12(10):793-800. doi: 10.1016/j.joca.2004.06.012. PMID 15450529
- [Background] De Mattei M, Varani K, Masieri FF, Pellati A, Ongaro A, Fini M, Cadossi R, Vincenzi F, Borea PA, Caruso A. Adenosine analogs and electromagnetic fields inhibit prostaglandin E2 release in bovine synovial fibroblasts. Osteoarthritis Cartilage. 2009 Feb;17(2):252-62. doi: 10.1016/j.joca.2008.06.002. Epub 2008 Jul 18. PMID 18640059
- [Background] Durmus A, Cakmak A, Disci R, Muslumanoglu L. The efficiency of electromagnetic field treatment in Complex Regional Pain Syndrome Type I. Disabil Rehabil. 2004 May 6;26(9):537-45. doi: 10.1080/09638280410001683155. PMID 15204461
- [Background] Fini M, Giavaresi G, Torricelli P, Cavani F, Setti S, Cane V, Giardino R. Pulsed electromagnetic fields reduce knee osteoarthritic lesion progression in the aged Dunkin Hartley guinea pig. J Orthop Res. 2005 Jul;23(4):899-908. doi: 10.1016/j.orthres.2005.01.008. Epub 2005 Mar 17. PMID 16023006
- [Background] Fini M, Torricelli P, Giavaresi G, Aldini NN, Cavani F, Setti S, Nicolini A, Carpi A, Giardino R. Effect of pulsed electromagnetic field stimulation on knee cartilage, subchondral and epyphiseal trabecular bone of aged Dunkin Hartley guinea pigs. Biomed Pharmacother. 2008 Dec;62(10):709-15. doi: 10.1016/j.biopha.2007.03.001. Epub 2007 Apr 3. PMID 17459652
- [Background] Gobbi A, Lad D, Petrera M, Karnatzikos G. Symptomatic Early Osteoarthritis of the Knee Treated With Pulsed Electromagnetic Fields: Two-Year Follow-up. Cartilage. 2014 Apr;5(2):78-85. doi: 10.1177/1947603513515904. PMID 26069687
- [Background] Comertoglu I, Gunes S, Elhan AH, Ustuner E, Kutlay S, Kucukdeveci AA. Effectiveness of pulsed electromagnetic field therapy in the management of complex regional pain syndrome type 1: A randomized-controlled trial. Turk J Phys Med Rehabil. 2022 Mar 1;68(1):107-116. doi: 10.5606/tftrd.2022.9074. eCollection 2022 Mar. PMID 35949961
- [Background] Marcheggiani Muccioli GM, Grassi A, Setti S, Filardo G, Zambelli L, Bonanzinga T, Rimondi E, Busacca M, Zaffagnini S. Conservative treatment of spontaneous osteonecrosis of the knee in the early stage: pulsed electromagnetic fields therapy. Eur J Radiol. 2013 Mar;82(3):530-7. doi: 10.1016/j.ejrad.2012.11.011. Epub 2012 Dec 3. PMID 23219192
- [Background] Moretti B, Notarnicola A, Moretti L, Setti S, De Terlizzi F, Pesce V, Patella V. I-ONE therapy in patients undergoing total knee arthroplasty: a prospective, randomized and controlled study. BMC Musculoskelet Disord. 2012 Jun 6;13:88. doi: 10.1186/1471-2474-13-88. PMID 22672794
- [Background] Notarnicola A, Covelli I, Moretti L, Setti S, De Terlizzi F, Moretti B. Predictors of responsiveness to biostimulation treatments (PEMFs and/or shockwaves) in patients with complex regional pain syndrome type I of the ankle. J Biol Regul Homeost Agents. 2021 May-Jun;35(3):1087-1095. doi: 10.23812/21-122-L. No abstract available. PMID 34155875
- [Background] Osti L, Buono AD, Maffulli N. Pulsed electromagnetic fields after rotator cuff repair: a randomized, controlled study. Orthopedics. 2015 Mar;38(3):e223-8. doi: 10.3928/01477447-20150305-61. PMID 25760511
- [Background] Pagani S, Veronesi F, Aldini NN, Fini M. Complex Regional Pain Syndrome Type I, a Debilitating and Poorly Understood Syndrome. Possible Role for Pulsed Electromagnetic Fields: A Narrative Review. Pain Physician. 2017 Sep;20(6):E807-E822. PMID 28934787
- [Background] Servodio Iammarrone C, Cadossi M, Sambri A, Grosso E, Corrado B, Servodio Iammarrone F. Is there a role of pulsed electromagnetic fields in management of patellofemoral pain syndrome? Randomized controlled study at one year follow-up. Bioelectromagnetics. 2016 Feb;37(2):81-8. doi: 10.1002/bem.21953. Epub 2016 Jan 12. PMID 26756278
- [Background] Smart KM, Wand BM, O'Connell NE. Physiotherapy for pain and disability in adults with complex regional pain syndrome (CRPS) types I and II. Cochrane Database Syst Rev. 2016 Feb 24;2(2):CD010853. doi: 10.1002/14651858.CD010853.pub2. PMID 26905470
- [Background] Ugras AA, Kural C, Kural A, Demirez F, Koldas M, Cetinus E. Which is more important after total knee arthroplasty: Local inflammatory response or systemic inflammatory response? Knee. 2011 Mar;18(2):113-6. doi: 10.1016/j.knee.2010.03.004. Epub 2010 May 14. PMID 20466551
- [Background] Varani K, De Mattei M, Vincenzi F, Gessi S, Merighi S, Pellati A, Ongaro A, Caruso A, Cadossi R, Borea PA. Characterization of adenosine receptors in bovine chondrocytes and fibroblast-like synoviocytes exposed to low frequency low energy pulsed electromagnetic fields. Osteoarthritis Cartilage. 2008 Mar;16(3):292-304. doi: 10.1016/j.joca.2007.07.004. Epub 2007 Aug 16. PMID 17698373
- [Background] Varani K, Gessi S, Merighi S, Iannotta V, Cattabriga E, Spisani S, Cadossi R, Borea PA. Effect of low frequency electromagnetic fields on A2A adenosine receptors in human neutrophils. Br J Pharmacol. 2002 May;136(1):57-66. doi: 10.1038/sj.bjp.0704695. PMID 11976268
- [Background] Veronesi F, Cadossi M, Giavaresi G, Martini L, Setti S, Buda R, Giannini S, Fini M. Pulsed electromagnetic fields combined with a collagenous scaffold and bone marrow concentrate enhance osteochondral regeneration: an in vivo study. BMC Musculoskelet Disord. 2015 Sep 2;16:233. doi: 10.1186/s12891-015-0683-2. PMID 26328626
- [Background] Veronesi F, Fini M, Giavaresi G, Ongaro A, De Mattei M, Pellati A, Setti S, Tschon M. Experimentally induced cartilage degeneration treated by pulsed electromagnetic field stimulation; an in vitro study on bovine cartilage. BMC Musculoskelet Disord. 2015 Oct 20;16:308. doi: 10.1186/s12891-015-0760-6. PMID 26480822
- [Background] Kotiuk V, Burianov O, Kostrub O, Khimion L, Zasadnyuk I. The impact of mirror therapy on body schema perception in patients with complex regional pain syndrome after distal radius fractures. Br J Pain. 2019 Feb;13(1):35-42. doi: 10.1177/2049463718782544. Epub 2018 Jun 13. PMID 30671237
- [Background] Vincenzi F, Targa M, Corciulo C, Gessi S, Merighi S, Setti S, Cadossi R, Goldring MB, Borea PA, Varani K. Pulsed electromagnetic fields increased the anti-inflammatory effect of A(2)A and A(3) adenosine receptors in human T/C-28a2 chondrocytes and hFOB 1.19 osteoblasts. PLoS One. 2013 May 31;8(5):e65561. doi: 10.1371/journal.pone.0065561. Print 2013. PMID 23741498
- [Background] Zorzi C, Dall'Oca C, Cadossi R, Setti S. Effects of pulsed electromagnetic fields on patients' recovery after arthroscopic surgery: prospective, randomized and double-blind study. Knee Surg Sports Traumatol Arthrosc. 2007 Jul;15(7):830-4. doi: 10.1007/s00167-007-0298-8. Epub 2007 Feb 28. PMID 17333120